CLINICAL TRIAL: NCT00501631
Title: Efficacy and Safety of VIVITROL® in Adults Completing Inpatient Treatment for Alcohol Dependence
Brief Title: ALK21-014: Efficacy and Safety of Medisorb® Naltrexone (VIVITROL®) After Enforced Abstinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK21-014
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Alcohol Dependence
Keywords: Addiction; Alcoholism; Inpatient detoxification
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIVITROL 380 mg (Active Comparator): Administered via intramuscular (IM) injection once every 4 weeks.
  Interventions: Drug: VIVITROL 380 mg
- Placebo for VIVITROL 380 mg (Placebo Comparator): Administered via IM injection once every 4 weeks.
  Interventions: Drug: Placebo for VIVITROL 380 mg

INTERVENTIONS:
Drug: VIVITROL 380 mg — Administered via IM injection once every 4 weeks.
  Other Names: naltrexone for extended-release injectable suspension; Medisorb naltrexone
  Arms: VIVITROL 380 mg
Drug: Placebo for VIVITROL 380 mg — Administered via IM injection once every 4 weeks.
  Arms: Placebo for VIVITROL 380 mg

SUMMARY:
VIVITROL is indicated for the treatment of alcohol dependence in patients who are able to abstain from alcohol in an outpatient setting prior to initiation of treatment with VIVITROL. This Phase 3B trial was designed to evaluate the efficacy and safety of VIVITROL versus placebo. Injections were administered to patients in whom abstinence was enforced by a period of inpatient hospitalization of 7 to 21 days.

DETAILED DESCRIPTION:
The study consisted of 2 parts, Part A and Part B. Part A was a double-blind, placebo-controlled assessment of safety and efficacy of VIVITROL versus placebo for 3 months. Part B was an open-label extension to assess longer-term safety, durability of effect, and health economics of VIVITROL when administered for up to 9 additional months.

ELIGIBILITY:
Primary Inclusion Criteria:

* Current diagnosis of alcohol dependence, meeting at least 5 of DSM-IV criteria
* Expected to complete inpatient treatment for alcohol dependence within 24 hours of randomization
* Must have 7-21 days, inclusive, of inpatient treatment for alcohol dependence prior to first dose
* Negative urine toxicological screen for opioids on the day of randomization
* Women of childbearing potential must agree to use an approved method of contraception for the study duration

Primary Exclusion Criteria:

* Pregnancy or lactation
* Evidence of hepatic failure including: ascites, bilirubin >10% above upper limit of normal and/or esophageal variceal disease
* Current dependence (within the past year) to benzodiazepines, opioids or cocaine by DSM-IV criteria
* Use of any opioids and/or methadone within 14 days prior to the screening visit, or subjects likely to require opioid therapy during the study period
* Use of oral naltrexone, acamprosate, or disulfiram within 14 days prior to screening
* Known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or PLG
* Parole, probation, or pending legal proceedings having the potential for incarceration during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- VIVITROL 380 mg: Arm includes all subjects who received at least 1 injection of VIVITROL. After successfully completing screening subjects were administered VIVITROL 380 mg by intramuscular (IM) injection every 4 weeks for a total of 3 injections. Randomization was 1:1 (VIVITROL:placebo) and stratified by site.
- Placebo for VIVITROL 380 mg: All subjects who received at least 1 injection of Placebo for VIVITROL. Arm includes all subjects who received at least 1 injection of placebo. After successfully completing screening subjects were administered placebo by intramuscular (IM) injection every 4 weeks for a total of 3 injections. Randomization was 1:1 (VIVITROL:placebo) and stratified by site.
Period: Part A (Double-blind Period)
Arm/Group | VIVITROL 380 mg | Placebo for VIVITROL 380 mg
Started | 152 | 148
Completed | 90 | 99
Not Completed | 62 | 49
Period: Part B (Open-label Period)
Arm/Group | VIVITROL 380 mg | Placebo for VIVITROL 380 mg
Started | 90 | 99
Completed | 37 | 48
Not Completed | 53 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIVITROL 380 mg | Placebo for VIVITROL 380 mg | Total
Number analyzed (Participants) | 152 | 148 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 152 | 148 | 300
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.5) | 46.1 (8.3) | 45.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 119 | 121 | 240
Region of Enrollment [Number; unit: participants]
  Germany | 142 | 138 | 280
  Austria | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percentage of Participants by Heavy Drinking Rate
Description: Cumulative percentage (%) of subjects reporting heavy drinking by category reflecting the various cut-offs for percentage of days that were heavy drinking days. A "heavy drinking day" was defined as 4 or more alcohol drinks in 1 day for women, and 5 or more alcohol drinks in 1 day for men. The Timeline Follow-Back (TLFB) method (Sobell & Sobell: Humana Press, 1992) was utilized to collect subjects' daily drinking information (ie, the number of drinks consumed per day per subject which was retrospectively recalled and recorded in a diary).
Time Frame: up to 12 weeks
Population: The primary endpoint is based on percentage rate of heavy drinking days during the double-blind treatment period as per protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Vivitrol | Placebo
Number analyzed (Participants) | 152 | 148
percentage of participants
  0% Heavy Drinking Days | 40.8 | 47.3
  <= 10% Heavy Drinking Days | 59.2 | 59.5
  <= 20% Heavy Drinking Days | 65.8 | 72.3
  <= 30% Heavy Drinking Days | 74.3 | 79.1
  <= 40% Heavy Drinking Days | 80.9 | 83.1
  <= 50% Heavy Drinking Days | 83.6 | 85.1
  <= 60% Heavy Drinking Days | 84.9 | 87.2
  <= 70% Heavy Drinking Days | 90.1 | 89.9
  <= 80% Heavy Drinking Days | 93.4 | 94.6
  <= 90% Heavy Drinking Days | 97.4 | 98.6
  <= 100% Heavy Drinking Days | 100.0 | 100.0
Statistical Analysis 1: Comparison: Vivitrol vs Placebo; The null hypothesis that there is no difference between two treatment groups (i.e. Placebo and Vivitrol) was tested using a two-sided Van der Waerden test. Response profiles were tabulated as a cumulative percent of subjects at each decile of percent heavy drinking days; Test type: Superiority or Other; p = 0.336, Van der Waerden test

2. Secondary Outcome: Longer-term Safety of VIVITROL
Description: Number of subjects reporting at least 1 treatment-emergent adverse event (TEAE) while on study.
Time Frame: up to 1 year
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Time Frame: AE collection began after a subject signed the informed consent form and continued until 30 days after the last dose of study drug was administered.
Description: All volunteered, elicited, and observed AEs were recorded on the AE CRFs.
Arm/Group | VIVITROL 380 mg (Double-blind Period) | Placebo for VIVITROL 380 mg (Double-blind Period)
Serious Adverse Events (participants affected / at risk) | 29/152 | 27/148
Other Adverse Events (participants affected / at risk) | 135/152 | 133/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIVITROL 380 mg (Double-blind Period) (N=152) | Placebo for VIVITROL 380 mg (Double-blind Period) (N=148)
Alcoholism (Psychiatric disorders) | 16 | 20
Suicidal ideation (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 1
Bereavement reaction (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 0 | 1
Psychosomatic disease (Psychiatric disorders) | 1 | 0
Somnolence (Psychiatric disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Injection site abscess (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0
Tibia fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Alcoholic seizure (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alcohol detoxification (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIVITROL 380 mg (Double-blind Period) (N=152) | Placebo for VIVITROL 380 mg (Double-blind Period) (N=148)
Injection site pain (General disorders) | 54 | 59
Fatigue (General disorders) | 15 | 5
Injection site induration (General disorders) | 7 | 3
Influenza like illness (General disorders) | 5 | 3
Alcoholism (Psychiatric disorders) | 25 | 40
Sleep disorder (Psychiatric disorders) | 8 | 10
Depression (Psychiatric disorders) | 9 | 7
Depressed mood (Psychiatric disorders) | 7 | 3
Headache (Nervous system disorders) | 25 | 25
Dizziness (Nervous system disorders) | 11 | 4
Nasopharyngitis (Infections and infestations) | 18 | 20
Nausea (Gastrointestinal disorders) | 20 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Toothache (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Hypertension (Vascular disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual Investigator may publish results without written agreement from Alkermes. Should an Investigator wish to publish or present the data at a meeting, a copy of the manuscript or abstract must be provided to the Sponsor at least 30 days prior to the submission for review and approval. Any revisions will be negotiated in good faith by the Investigator and Sponsor.